CLINICAL TRIAL: NCT01338337
Title: Multicentre, Open-label, Randomized Phase II Study of Vidaza (Azacitidine) Versus Support Treatment in Patients With Low Risk Myelodysplastic Syndrome (Low and Intermediate-1 International Prognostic Scoring System(IPSS )) Without the 5q Deletion and Transfusion Dependent Anaemia
Brief Title: Study of Vidaza (Azacitidine) Versus Support Treatment in Patients With Low Risk Myelodysplastic Syndrome (Low and Intermediate-1 IPSS) Without the 5q Deletion and Transfusion Dependent Anaemia
Acronym: ABRAZA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asociación Andaluza de Hematología y Hemoterapia (Other)
Responsible Party: Principal Investigator, Joaquin Sanchez, MD. Ph D Hematologist, Asociación Andaluza de Hematología y Hemoterapia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABRAZA
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Low risk International Prognostic Scoring System (IPSS) (0 or Int-1); Patients who have not responded to previous treatment with erythropoietin (EPO); Eastern Cooperative Oncology Group (ECOG) score ≤ 3
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Support treatment (No Intervention): Transfusional support will be applied for symptomatic anaemia using clinical discretion and chelation therapy when ferritin is ≥ 1000 μgr/ml with the chelating agents allowed.
- Azacitidine (Experimental): Azacitidine 75 mg/m2, for 5 days of each 20 day cycle. Transfusional support will be applied for symptomatic anaemia using clinical discretion and chelation therapy when ferritin is ≥ 1000 μgr/ml with the chelating agents allowed
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 75 mg/m2, for 5 days of each 20 day cycle. Transfusional support will be applied for symptomatic anaemia using clinical discretion and chelation therapy when ferritin is ≥ 1000 μgr/ml with the chelating agents allowed
  Arms: Azacitidine

SUMMARY:
Primary Outcome Measures:

• To evaluate the efficacy of treatment with Azacitidine in patients with transfusion-dependent, low risk International Prognostic Scoring System (IPSS) 0 int-1, Myelodysplastic Syndrome (MDS) without chromosome 5 (5q) deletion. The main objective will be based on the erythroid haematologic response according to International Working Group (IWG) 2006 criteria.

Secondary Outcome Measures:

* Haematologic response, bases on the following parameters: platelets, and neutrophils according to International Working Group (IWG) Criteria.
* Medullary and cytogenetic response according to International Working Group (IWG) 2006 criteria.
* The effect of treatment response on quality of life, through the Functional Assessment of Cancer Therapy-Anemia (FACT-an) questionnaire.
* Overall survival, Event-Free Survival and the Acute Leukaemia Transformation Rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age.
2. Patients who agree to take part in the study must understand the informed consent and sign it voluntarily.
3. Patients must be able to comply with all the programmed visits and other study requirements.
4. Patients with low risk International Prognostic Scoring System (IPSS 0 or Int-1) myelodysplastic syndrome (MDS) without chromosome 5 (5q) deletion and anaemia with transfusion needs. Transfusion dependence is defined as at least 2 units of erythrocyte concentrate (EC) during the 8 weeks prior to inclusion in the study, and symptomatic anaemia, defined by a haemoglobin value ≤9.0 gr/dl.
5. Patients who have not responded to previous treatment with erythropoietin (EPO): With a response profile based on basal erythropoietin (EPO) levels of > 250 u/L, with no response alter 12 weeks of treatment at maximum doses (60.000 U or 250 µg darbepoetin (DAB), in combination with Granulocyte colony-stimulating factor (G-CSF) in cases of refractory anaemia with ringed sideroblasts (RARS)) , or with loss of the response obtained after an initial optimum response.
6. Patients who are not candidates for intensive chemotherapy and transplant modalities.
7. Patients with an Eastern Cooperative Oncology Group (ECOG) score ≤ 3
8. Women of child-bearing age and heterosexual men whose partner is of child-bearing age, must undertake to use an effective contraceptive method for the duration of the treatment and for at least 3 months alter is has finalised.

Exclusion Criteria:

1. The presence of a psychiatric or medical disease which prevents the patient from signing of the informed consent.
2. Human immunodeficiency virus (HIV) Seropositive, hepatitis B antigen (AgVHB) positive or hepatitis C virus (HCV) polymerase chain reaction (PCR) positive.
3. Pregnant or nursing women.
4. Uncontrolled intercurrent disease: Active infection requiring parenteral antibiotics, Symptomatic chronic heart failure (New York Heart Association (NYHA) class III or IV), Instable angina pectoris, or Another neoplasia apart from his myelodysplastic syndromes (MDS).
5. Have been treated with demethylating drugs at any moment prior to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Erythroid haematologic response | Approximately the primary outcome is measured on days 0, 252 and 504 (basal, cycle 9 and 18 (each cicle has 28 days +/-3 days))
  To evaluate the efficacy of treatment with Azacitidine in patients with transfusion-dependent, low risk International Prognostic Scoring System (IPSS) 0 or int-1, Myelodysplastic Syndrome (MDS) without chromosome 5 (5q) deletion. The main objective will be based on the erythroid haematologic response according to International Working Group (IWG) 2006 criteria.

SECONDARY OUTCOMES:
Haematologic response | The secondary outcome is measured on days 0, 28, 56, 84, 112, 140, 168, 196, 224, 252, 280, 308, 336, 364, 392, 420, 448, 476 and 504 (the measurement is performed at basal line and in every cycle (every 28 days +/-3 days) up to a maximum of 18 cycles).
  Haematologic response, bases on the following parameters: platelets, and neutrophils according to International Working Group (IWG) Criteria.
Medullary and cytogenetic response | Approximately this secondary outcome is measured on days 252 and 504 (basal, cycle 9 and 18 (each cicle has 28 days +/-3 days)).
  Medullary and cytogenetic response according to International Working Group (IWG) 2006 criteria.
Quality of life | Approximately this secondary outcome is measured on days 252 and 504 (basal, cycle 9 and 18 (each cicle has 28 days +/-3 days)).
  The effect of treatment response on quality of life, through the Functional Assessment of Cancer Therapy-Anemia (FACT-An) questionnaire.
Overall survival | The secondary outcome is measured from basal line until day 504 (average of days for 18 cycles), or until progresion, or until exitus... (from basal line until the end of the study)
  Overall survival
Event-Free Survival | The secondary outcome is measured from basal line until day 504 (average of days for 18 cycles), or until progresion, or until exitus... (from basal line until the end of the study)
  Event-Free Survival
Acute Leukaemia Transformation Rate | The secondary outcome is measured from basal line until day 504 (average of days for 18 cycles), or until progresion, or until exitus... (from basal line until the end of the study)
  Acute Leukaemia Transformation Rate

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Reina Sofía, Servicio de Hematología, Córdoba, Cordoba
  - Hospital General de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario San Cecilio, Granada, Granada
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Virgen de Valme, Seville, Sevilla